CLINICAL TRIAL: NCT02082054
Title: A Phase 2, Double-Blind, Parallel-Group, Dose-Ranging Study Evaluating Safety/ Efficacy Atropine Doses With Pseudoephedrine and Chlorpheniramine in SAR Patients 12 Years of Age and Older
Brief Title: StahistRx Phase 2, Five-arm, Parallel Group, Active vs Active, Double-blind Study
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Magna Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MAGNA2014-001
Record Dates: First submitted 2014-02-26; First posted 2014-03-10 (Estimated); Last update posted 2014-05-30 (Estimated); Status verified 2014-02

CONDITIONS: Rhinitis, Seasonal, Allergic
Keywords: rhinitis; seasonal; allergic
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal; Rhinitis | interventions — Proto-Oncogene Proteins c-raf; Pseudoephedrine; Chlorpheniramine; Atropine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- PSE 120 mg, CM 8 mg, Atr 0.36 mg (Experimental): Pseudoephedrine 120 mg,chlorpheniramine 8 mg, atropine 0.36 mg tablet dosed BID for 7.5 days
  Interventions: Drug: PSE 120 mg, CM 8 mg, Atr 0.36 mg
- PSE 120 mg, CM 8 mg, Atr 0.24 mg (Experimental): Pseudoephedrine 120 mg, chlorpheniramine 8 mg, atropine 0.24 mg tablets dosed BID for 7.5 days
  Interventions: Drug: PSE 120 mg, CM 8 mg, Atr 0.24 mg
- PSE 120 mg, CM 8 mg, Atr 0.12 mg (Experimental): Pseudoephedrine 120 mg, chlorpheniramine 8 mg, atropine 0.12 dosed BID for 7.5 days
  Interventions: Drug: PSE 120 mg, CM 8 mg, Atr 0.12 mg
- PSE 120 mg, CM 8 mg (Active Comparator): Pseudoephedrine 120 mg, chlorpheniramine 8 mg white, scored, tablets with "M27" on scored side and plain on the other side
  Interventions: Drug: PSE 120 mg, CM 8 mg
- Atropine 0.24 mg (Experimental): Atropine 0.24 mg tablets dosed BID for 7.5 days
  Interventions: Drug: Atropine 0.24 mg

INTERVENTIONS:
Drug: PSE 120 mg, CM 8 mg, Atr 0.36 mg — Pseudoephedrine 120 mg, chlorpheniramine 8 mg, atropine 0.36 mg white, scored, tablets with "M27" on scored side and plain on the other side
  Other Names: Pseudoephedrine, chlorpheniramine (Chlor-Trimeton), atropine
  Arms: PSE 120 mg, CM 8 mg, Atr 0.36 mg
Drug: PSE 120 mg, CM 8 mg, Atr 0.24 mg — Pseudoephedrine 120 mg, chlorpheniramine 8 mg, atropine 0.24 mg white, scored, tablets with "M27" on scored side and plain on the other side
  Other Names: Pseudoephedrine, chlorpheniramine (Chlor-Trimeton), atropine
  Arms: PSE 120 mg, CM 8 mg, Atr 0.24 mg
Drug: PSE 120 mg, CM 8 mg, Atr 0.12 mg — Pseudoephedrine 120 mg, chlorpheniramine 8 mg, atropine 0.12 mg white, scored, tablets with "M27" on scored side and plain on the other side
  Other Names: Pseudoephedrine, chlorpheniramine (Chlor-Trimeton), atropine
  Arms: PSE 120 mg, CM 8 mg, Atr 0.12 mg
Drug: PSE 120 mg, CM 8 mg — Pseudoephedrine 120 mg, chlorpheniramine 8 mg tablets dosed BID
  Other Names: Pseudoephedrine, chlorpheniramine (Chlor-Trimeton)
  Arms: PSE 120 mg, CM 8 mg
Drug: Atropine 0.24 mg — Atropine sulfate 0.24 mg white, scored, tablets with "M27" on scored side and plain on the other side
  Other Names: atropine sulfate
  Arms: Atropine 0.24 mg

SUMMARY:
This active vs active comparative trial will evaluate the safety and efficacy of incremental doses of atropine in combination with pseudoephedrine 120 mg/chlorpheniramine 8 mg in adult patients with a history of seasonal allergic rhinitis. Hypotheses are defined by total nasal symptom scores (TNSS) recorded by subjects in diaries where efficacy will be established by statistical significance where p < 0.05.

DETAILED DESCRIPTION:
Actives in each of the five study arms:

Pseudoephedrine 120 mg/Chlorpheniramine 8 mg/Atropine 0.36 mg Pseudoephedrine 120 mg/Chlorpheniramine 8 mg/Atropine 0.24 mg Pseudoephedrine 120 mg/Chlorpheniramine 8 mg/Atropine 0.12 mg Pseudoephedrine 120 mg/Chlorpheniramine 8 mg Atropine 0.24 mg

ELIGIBILITY:
Inclusion Criteria:

1. Male and females of any ethnic group between 12 and 60 years of age.
2. History of moderate to severe SAR for at least two years; defined as having a score of 2 or more on a 0-3 point scale
3. Documentation of sensitivity will be obtained from medical records or positive skin testing or in vitro specific IgE test.
4. Have a TNSS score of 6 with at least an average of 2.0 in the rhinorrhea sub-score during the placebo-run in phase.
5. Is a non-pregnant, non-lactating female who is postmenopausal, naturally or surgically sterile, or who agree to use effective contraceptive methods throughout the course of the study.
6. If female of childbearing potential, must agree to use listed acceptable birth control methods...
7. If female of childbearing potential, has a negative urine human chorionic gonadotropin (hCG) pregnancy test at screening
8. Is able to swallow whole tablets of orally administered medication
9. Is able to understand and provide signed informed consent

Exclusion Criteria:

1. Has asthma requiring corticosteroid treatment
2. Is currently undergoing chronic or intermittent use of inhaled, oral, intramuscular, intravenous, and/or potent or super potent topical corticosteroids
3. Has taken any of the following medications in the indicated time period prior to study enrolment:

   * Intranasal, opthalmic, or systemic corticosteroids (1 month)
   * Intranasal cromolyn (2 weeks)
   * Intranasal or systemic decongestants (3 days)
   * Intranasal or systemic antihistamines (7 days) or leukotriene inhibitors (7 days)
4. Documented evidence of acute or significant chronic sinusitis, as determined by the individual investigator
5. Has a history of allergic reaction to or known sensitivity to the active or inactive ingredients in the investigational products used in this study
6. Chronic use of concomitant medications (e.g., tricyclic antidepressants) that would affect assessment of the effectiveness of the study medication
7. Rhinitis medicamentosa
8. A history of glaucoma
9. Has known or suspected pregnancy, planned pregnancy, or lactation (for female patients)
10. Is currently receiving immunotherapy, unless at stable maintenance dose for at least 1 month.
11. Presence of a medical condition that might interfere with treatment evaluation or require a change in therapy.
12. Plans to travel outside the study area for a substantial portion of the study period
13. Has a history in the last 2 years or current evidence of abuse of illicit drugs, prescription medications, or alcohol that, in the opinion of the Investigator, would interfere with adherence to study requirements.
14. Has exposure to any investigational agent within 30 days prior to study entry.
15. Has clinically significant mental illness (to be determined by the Investigator)
16. Has a condition the Investigator believes would interfere with the ability to provide informed consent or comply with study instructions, or that might confound the interpretation of the study results or put the patient at undue risk

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 125 (Estimated)
Dates: Start 2014-03; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
Dose-ranging data for atropin | 7.5 days
  To provide dose-ranging data for atropine and select a dose of Atropine for Phase 3 clinical development using Total Nasal Symptom Score (TNSS) as the primary endpoint plus recording of adverse events

SECONDARY OUTCOMES:
Establish effect size for determining power and TNSS efficacy endpoint | 7.5 days
  To establish an effect size of a Pseudoephedrine 120 mg/Chlorpheniramine 8 mg/Atropine combination versus Pseudoephedrine 120 mg/Chlorpheniramine 8 mg to statistically power the pivotal phase of the study using TNSS as the primary endpoint

OTHER OUTCOMES:
Establish safety/efficacy and appropriate dosage interval of investigational formulas | 7.5 days
  1. Assess the instantaneous and reflective TNSS scores.
  2. To assess the effect of various doses of Atropine in combination with Pseudoephedrine 120 mg/Chlorpheniramine 8 mg on each of the four (4) individual components of the TNSS compared to Pseudoephedrine 120 mg/Chlorpheniramine 8 mg alone
  3. To assess if BID dosing is an appropriate dosing interval for the Pseudoephedrine/Chlorpheniramine/Atropine formulation
  4. To assess the effect of Atropine 0.24 mg alone on the change from baseline of each of the four (4) individual components of the TNSS
  5. To assess the safety and tolerability of Pseudoephedrine 120 mg/Chlorpheniramine 8 mg/Atropine combination products compared to Pseudoephedrine 120 mg/Chlorpheniramine 8 mg product as well as the safety and tolerability of atropine 0.24 mg administered twice/day.
  6. To assess the incidence and severity of drowsiness

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J Pollard, MD, Principal Investigator — Family Allergy and Asthma
Locations (4):
- United States (4):
  - Clinical Research Atlanta, Stockbridge, Georgia
  - Family Allergy and Asthma Institute, Louisville, Kentucky
  - National Allergy, Asthma & Urticaria Centers of Charleston, PA, Charleston, South Carolina
  - Central Texas Health Research, New Braunfels, Texas